CLINICAL TRIAL: NCT02920177
Title: Platelet-rich Plasma Versus Corticosteroid Injection for the Treatment of Femoroacetabular Impingement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Tariq Awan, Assistant Professor in Orthopaedic Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00104340
Record Dates: First submitted 2016-08-30; First posted 2016-09-30 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Femoroacetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- platelet-rich plasma (Experimental): platelet-rich plasma injection into the head-neck junction of the hip joint
  Interventions: Drug: platelet-rich plasma injection
- Kenalog 10 mg/mL Injectable Suspension (Active Comparator): corticosteroid injection into the head-neck junction of the hip joint
  Interventions: Drug: Kenalog 10 MG/ML Injectable Suspension

INTERVENTIONS:
Drug: platelet-rich plasma injection — platelet-rich plasma injection
  Other Names: PRP
  Arms: platelet-rich plasma
Drug: Kenalog 10 MG/ML Injectable Suspension — 4 mL corticosteroid injection
  Arms: Kenalog 10 mg/mL Injectable Suspension

SUMMARY:
The purpose of this study is to compare the clinical response of intra-articular platelet rich plasma (PRP) versus corticosteroid injection in patients affected by femoroacetabular impingement (FAI).

DETAILED DESCRIPTION:
This study will determine if PRP treatment of FAI improves (i) patient reported outcome scores and (ii) hip functional stability compared to standard corticosteroid treatment and if PRP treatment of FAI reduces (i) radiographic and (ii) biochemical markers of joint inflammation and cartilage degradation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic FAI
* Clinical and radiographic evidence of FAI
* Patients able to provide consent to study participation
* Completion of 6 weeks of physical therapy program

Exclusion Criteria:

* Established Osteoarthritis (Kellgren-Lawrence > 3)
* Minimum joint space > 2 mm as measured on AP radiograph
* Hip dysplasia (center edge angle < 20° on AP radiograph)
* Patients with clinically significant cardiovascular, renal, hepatic, endocrine disease, cancer or diabetes
* Patients with ongoing infection including HIV and Hepatitis
* Patient with history of osteomyelitis/septic arthritis
* Anticoagulation therapy
* Patients who are pregnant or breast feeding
* Patients with systemic, rheumatic or inflammatory disease of the knee or chondrocalcinosis, hemochromatosis, inflammatory arthritis, arthropathy of the knee associated with juxta-articular Paget's disease of the femur or tibia, hemophilic arthropathy, infectious arthritis, Charcot's knee joint, villonodular synovitis, and synovial chondromatosis
* Patients taking immunosuppressant medication
* Patients with abnormal hematology or serum chemistry lab results
* Patients receiving injection to treatment knee within 2 months of study enrollment
* BMI greater than 35 or less than 20

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tariq M Awan, DO, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Platelet-rich Plasma | Kenalog 10 mg/mL Injectable Suspension
Started | 2 | 2
Completed | 0 | 0
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platelet-rich Plasma | Kenalog 10 mg/mL Injectable Suspension | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Kellgren-Lawrence classification scores [Mean (Full Range); unit: score on a scale] — Kellgren Lawrence grading system will be utilized analyzing pre-treatment and post-treatment radiographs of the knee. Grading is from 1 to 4 with 1 being minimal to mild disease and 4 being end stage joint disease.
  score on a scale | 1 [0 to 1] | 2 [1 to 2] | 1 [0 to 2]
Pain as measured by Visual Analog Scale (VAS) [Mean (Full Range); unit: score on a scale] — VAS score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
  score on a scale | 53.5 [50 to 57] | 53 [40 to 66] | 53.25 [40 to 66]
Serum Biomarkers [Mean (Full Range); unit: pg/mL]
  IFN-g | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected
  IL-6 | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected
  MCP-1 | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected
  MIP-1b | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected
  IL-1b | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected
  TNF-alpha | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected
  high-sensitivity CRP | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected
  COMP | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected | NA [NA to NA] — Samples were collected, but never analyzed as the study was terminated before any outcome measure data could be collected
HOOS Hip Survey [Mean (Full Range); unit: score on a scale] — Hip Disability and Osteoarthritis Outcome Score (HOOS) is a hip-specific patient-reported outcome measure that has 5 subscales. Each subscale is scored separately and ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
  score on a scale
    HOOS Symptom Score | 57.5 [40 to 75] | 47.5 [45 to 50] | 52.5 [40 to 75]
    HOOS Activities of Daily Living | 84 [72 to 96] | 61.5 [59 to 64] | 72.75 [59 to 96]
    HOOS Sports and Recreation Score | 84.5 [81 to 88] | 45.5 [25 to 66] | 65 [25 to 88]
    HOOS Quality of Life Score | 53.5 [44 to 63] | 23 [19 to 27] | 38.25 [19 to 63]
    HOOS Pain Score | 72.5 [60 to 85] | 50 [45 to 55] | 61.25 [45 to 85]
Patient Reported Outcome Measurement Information System (PROMIS) Global Health Scale [Mean (Full Range); unit: score on a scale] — Global physical health measures overall physical health, physical function, pain and fatigue. Physical global health scores range from 0 - 100, and higher scores indicate better physical health.
  Global mental health measures mental health, quality of life, satisfaction with social activities and emotional problems. Global mental health scores range from 0 - 100, and higher scores indicate better mental health.
  score on a scale
    Physical Health | 16 [15 to 17] | 16 [16 to 16] | 16 [15 to 17]
    Mental Health | 14.5 [13 to 16] | 13 [12 to 14] | 13.75 [12 to 16]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pain Score on the Visual Analog Scale
Description: VAS score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Time Frame: 12 months
Population: No twelve month data was collected because none of the endpoints were reached. All participants left the study before the 6 month follow up.
Arm/Group | Platelet-rich Plasma | Kenalog 10 mg/mL Injectable Suspension
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Hip Disability and Osteoarthritis Outcome Score (HOOS), Western Ontario and McMaster Universities Arthritis Index (WOMAC), Calculated as a Sub-score of the HOOS
Description: Measure Description: Hip Disability and Osteoarthritis Outcome Score (HOOS) is a hip-specific patient-reported outcome measure that has 5 subscales. Each subscale is score separately and ranges from 0-100, 100 = no disability, therefore higher values indicate a better outcome.
  The WOMAC (Western Ontario and McMaster Universities) index is used to assess patients with osteoarthritis of the hip or knee and contains 24 questions, targeting areas of pain, stiffness and physical function. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). WOMAC total is the sum of the three components and it ranges from 0 to 96 points, being 96 the worst outcome.
  The questions that are included in the WOMAC are a subgroup of questions that are included in the HOOS, so because of this the HOOS survey can also be used to calculate the WOMAC score for patients.
Time Frame: 12 months
Population: as for outcome 1
Arm/Group | Platelet-rich Plasma | Kenalog 10 mg/mL Injectable Suspension
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Patient Reported Outcome Measurement Information System (PROMIS) Global Health Scale
Description: Global mental health measures mental health, quality of life, satisfaction with social activities and emotional problems. Global mental health scores range from 0 - 100, and higher scores indicate better mental health.
  Global physical health measures overall physical health, physical function, pain and fatigue. Physical global health scores range from 0 - 100, and higher scores indicate better physical health.
Time Frame: 12 months
Population: as for outcome 1
Arm/Group | Platelet-rich Plasma | Kenalog 10 mg/mL Injectable Suspension
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Serum Biomarker Analysis: IFN-g, IL-6, MCP-1, MIP-1b, IL-1b, TNF-alpha, Highly Sensitive CRP, COMP.
Time Frame: 12 months
Population: as for outcome 1
Arm/Group | Platelet-rich Plasma | Kenalog 10 mg/mL Injectable Suspension
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Kellgren-Lawrence Classification Scores
Description: Calculated from anterior-posterior (AP) pelvis radiographs. Kellgren Lawrence grading system was intended to be utilized analyzing pre-treatment and post-treatment radiographs of the knee. Grading is from 1 to 4 with 1 being minimal to mild disease and 4 being end stage joint disease.
Time Frame: 12 months
Population: as for outcome 1
Arm/Group | Platelet-rich Plasma | Kenalog 10 mg/mL Injectable Suspension
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Platelet-rich Plasma | Kenalog 10 mg/mL Injectable Suspension
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Recruitment was supposed to take place in the first year, but was extended due to low enrollment. The study was terminated early due to an inability to enroll subjects. All participants left the study before outcome measure data could be collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT02920177/Prot_SAP_000.pdf